CLINICAL TRIAL: NCT01652157
Title: A Long-Term Prospective Observational Safety Study of the Incidence of and Risk Factors for Fibrosing Colonopathy in US Patients With Cystic Fibrosis Treated With Pancreatic Enzyme Replacement Therapy: A Harmonized Protocol Across Sponsors(The CF-FC Study)
Brief Title: Long-term Study in US Cystic Fibrosis Patients Receiving Digestive Enzyme Supplements to Assess Narrowing of the Large Intestine Causing Adverse Intestinal Symptoms (Fibrosing Colonopathy)
Status: Terminated | Type: Observational
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Collaborators: Cystic Fibrosis Foundation (Other); Digestive Care, Inc. (Industry); Nestle Health Science (Industry); VIVUS LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CFFC-OB-11
Record Dates: First submitted 2012-07-25; First posted 2012-07-27 (Estimated); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Fibrosing Colonopathy
Keywords: prospective; observational; pancreatic insufficiency; pancreatic enzyme replacement therapy; fibrosing colonopathy; patients with cystic fibrosis
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency | interventions — Pancrelipase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cystic fibrosis (CF) patients in the CF Patient Registry: Patients diagnosed with cystic fibrosis at participating sites who are providing data to the Cystic Fibrosis Patient Registry
  Interventions: Biological: ULTRESA; Biological: PANCREAZE; Biological: CREON; Biological: ZENPEP; Biological: other non-sponsor pancreatic enzyme replacement therapy; Biological: PERTZYE; Other: No pancreatic enzyme replacement therapy

INTERVENTIONS:
Biological: ULTRESA — pancreatic enzyme replacement therapy
  Other Names: pancrelipase
Biological: PANCREAZE — pancreatic enzyme replacement therapy
  Other Names: pancrelipase
Biological: CREON — pancreatic enzyme replacement therapy
  Other Names: pancrelipase
Biological: ZENPEP — pancreatic enzyme replacement therapy
  Other Names: pancrelipase
Biological: other non-sponsor pancreatic enzyme replacement therapy — pancreatic enzyme replacement therapy
  Other Names: pancrelipase
Biological: PERTZYE — pancreatic enzyme replacement therapy
  Other Names: pancrelipase
Other: No pancreatic enzyme replacement therapy — Cystic fibrosis patients in the cystic fibrosis registry not receiving any pancreatic enzyme replacement therapy (approximately 10%)

SUMMARY:
This is a long-term study in cystic fibrosis patients who are participating in the Cystic Fibrosis Patient Registry to assess the occurrence and risk factors for a rare bowel disorder called fibrosing colonopathy (narrowing of the large intestine). Patients will be followed at their regular clinical care visits over a 10-year period and approached if they develop symptoms of fibrosing colonopathy for collection and use of further detailed information.

DETAILED DESCRIPTION:
This is a prospective, observational, population-based cohort study in US cystic fibrosis patients participating in the Cystic Fibrosis Patient Registry in order to assess the incidence of and risk factors for fibrosing colonopathy. Cystic fibrosis (CF) patients participating in the registry from participating sites, as well as new CF patients enrolled in the registry at these sites over a 2-year period, will serve as the base study population (estimated to include 24,500-25,000 cystic fibrosis patients between the first patient encounter documented in the registry from any participating site and the 31st of July 2014). Cystic fibrosis patients in the base study population will be followed at their regular clinical care visits and, any patients presenting over a 10-year period with signs and symptoms of suspected fibrosing colonopathy, based on a prospective definition, will be approached to obtain a study-specific informed consent for collection of additional data outside the standard registry data collection form in order to augment surveillance. Data routinely collected via the standard CF registry will be used to determine exposure to any specific pancreatic enzyme replacement therapy and to assess potential risk factors for the outcome of confirmed fibrosing colonopathy. An independent adjudication panel will be utilized to validate the diagnosis of fibrosing colonopathy based on a prospective case definition as well as decision rules.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria for enrollment in the Base Study Population

* Diagnosed with cystic fibrosis,
* Enrolled in the Cystic Fibrosis Patient Registry
* Receiving medical care at a Cystic Fibrosis Foundation-accredited care center providing data to the Cystic Fibrosis Patient Registry

Exclusion Criteria:

* None

Ages: 0 Months to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cystic fibrosis patients who are active in the Cystic Fibrosis Patient Registry
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2012-07-31 (Actual); Primary Completion 2020-04-08 (Actual); Study Completion 2020-04-08 (Actual)

PRIMARY OUTCOMES:
Incidence rate of fibrosing colonopathy confirmed by an independent adjudication panel in patients receiving ZENPEP | up to 10 years
  Fibrosing colonopathy is confirmed by an independent adjudication panel based on prospectively defined criteria.
Incidence rate of fibrosing colonopathy confirmed by an independent adjudication panel in patients receiving ULTRESA | up to 10 years
  Fibrosing colonopathy is confirmed by an independent adjudication panel based on prospectively defined criteria.
Incidence rate of fibrosing colonopathy confirmed by an independent adjudication panel in patients receiving PERTZYE. | up to 10 years
  Fibrosing colonopathy is confirmed by an independent adjudication panel based on prospectively defined criteria.
Incidence rate of fibrosing colonopathy confirmed by an independent adjudication panel in patients receiving CREON | up to 10 years
  Fibrosing colonopathy is confirmed by an independent adjudication panel based on prospectively defined criteria.
Incidence rate of fibrosing colonopathy confirmed by an independent adjudication panel in patients receiving PANCREAZE | up to 10 years
  Fibrosing colonopathy is confirmed by an independent adjudication panel based on prospectively defined criteria.
Incidence rate of fibrosing colonopathy confirmed by an independent adjudication panel in patients not receiving pancreatic enzyme therapy. | up to 10 years
  Fibrosing colonopathy is confirmed by an independent adjudication panel based on prospectively defined criteria.
Incidence rate of fibrosing colonopathy confirmed by an independent adjudication panel in patients receiving non-sponsor pancreatic enzyme replacement therapy | up to 10 years
  Fibrosing colonopathy is confirmed by an independent adjudication panel based on prospectively defined criteria.

SECONDARY OUTCOMES:
Odds ratio (95% confidence interval) to quantify the association between possible risk factors and confirmed fibrosing colonopathy | up to 10 years
  Potential risk factors include demographics, medical history, and concurrent medications, including daily dosage and length of specific pancreatic enzyme replacement therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Craig Peterson, Study Director — VIVUS LLC
Locations (123):
- United States (123):
  - Children's Hospital of Alabama /ID# 78920, Birmingham, Alabama
  - Alaska Medical Center /ID# 79256, Anchorage, Alaska
  - Phoenix Children's Hospital /ID# 78906, Phoenix, Arizona
  - University of Arizona Cancer Center - North Campus /ID# 78939, Tucson, Arizona
  - Arkansas Children's Hospital /ID# 79265, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences /ID# 76785, Little Rock, Arkansas
  - Ucsd /Id# 105039, La Jolla, California
  - Loma Linda University /ID# 79237, Loma Linda, California
  - Miller Childrens Hospital /ID# 78896, Long Beach, California
  - Kaiser Permanente Regional Met /ID# 79235, Los Angeles, California
  - Usc /Id# 76793, Los Angeles, California
  - Children's Hosp and Res Ctr /ID# 79295, Oakland, California
  - Kaiser Permanente /ID# 78899, Oakland, California
  - UC Davis Comprehensive Cancer Center - Main /ID# 118935, Sacramento, California
  - California Pacific Medical Ctr /ID# 76775, San Francisco, California
  - Univ California, San Francisco /ID# 78925, San Francisco, California
  - Stanford University /ID# 95156, Stanford, California
  - Univ of Colorado Cancer Center /ID# 79277, Aurora, Colorado
  - National Jewish Health /ID# 76784, Denver, Colorado
  - CT Childrens Medical Ctr, US /ID# 78923, Hartford, Connecticut
  - Yale University /ID# 78940, New Haven, Connecticut
  - Nemours/Alfred duPont Hospital for Children /ID# 78945, Wilmington, Delaware
  - Children's National Medical Center /ID# 79373, Washington D.C., District of Columbia
  - Central FL Pulmonary Altamonte /ID# 76776, Altamonte Springs, Florida
  - University of Florida - Archer /ID# 76790, Gainesville, Florida
  - University of Florida - Archer /ID# 78928, Gainesville, Florida
  - Joe DiMaggio Children's Hospital at Memorial /ID# 79234, Hollywood, Florida
  - Nemour Child Clin FL, US /ID# 78898, Jacksonville, Florida
  - University of Miami, Miller School of Medicine /ID# 78927, Miami, Florida
  - Nemours Children's Clinic /ID# 78917, Orlando, Florida
  - Arnold Palmer Hosp Children /ID# 96075, Orlando, Florida
  - All Children's Hospital /ID# 79264, St. Petersburg, Florida
  - Emory University Hospital /ID# 79394, Atlanta, Georgia
  - Children's Healthcare of Atlanta - Ferry Rd /ID# 116275, Atlanta, Georgia
  - Georgia Regents University /ID# 79395, Augusta, Georgia
  - St Luke's Cystic Fibrosis Center of Idaho /ID# 79259, Boise, Idaho
  - Duplicate_Childrens Hospital of Chicago /ID# 79296, Chicago, Illinois
  - University of Chicago /ID# 78924, Chicago, Illinois
  - Loyola University Medical Ctr /ID# 76780, Maywood, Illinois
  - Advocate Lutheran Gen Children /ID# 76781, Park Ridge, Illinois
  - OSF Saint Francis Medical Ctr /ID# 78905, Peoria, Illinois
  - Lutheran Hospital of Indiana /ID# 79238, Fort Wayne, Indiana
  - Indiana University /ID# 121395, Indianapolis, Indiana
  - Indiana University /ID# 78903, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics /ID# 78921, Iowa City, Iowa
  - University of Kansas Health Sy /ID# 78929, Kansas City, Kansas
  - Via Christi Specialty Clinics /ID# 78946, Wichita, Kansas
  - Kentucky Clinic /ID# 78922, Lexington, Kentucky
  - University of Louisville /ID# 78926, Louisville, Kentucky
  - Tulane Univ /ID# 78916, New Orleans, Louisiana
  - Louisiana State Univ HSC /ID# 78943, Shreveport, Louisiana
  - MMP Women's Health /ID# 78894, Portland, Maine
  - Johns Hopkins University /ID# 78893, Baltimore, Maryland
  - Tufts-New England Medical Ctr /ID# 79254, Boston, Massachusetts
  - Massachusetts General Hospital /ID# 78895, Boston, Massachusetts
  - Boston Childrens Hospital /ID# 79276, Boston, Massachusetts
  - Baystate Medical Center /ID# 103437, Springfield, Massachusetts
  - UMass Memorial Medical Center /ID# 78954, Worcester, Massachusetts
  - University of Michigan Hospitals /ID# 99035, Ann Arbor, Michigan
  - Children's Hospital of MI /ID# 79278, Detroit, Michigan
  - Michigan State University /ID# 78950, East Lansing, Michigan
  - Helen DeVos Childrens Hospital /ID# 79397, Grand Rapids, Michigan
  - University of Minnesota /ID# 76791, Minneapolis, Minnesota
  - Univ of Mississippi Med Ctr,US /ID# 78934, Jackson, Mississippi
  - University of Missouri /ID# 109755, Columbia, Missouri
  - The Children's Mercy Hospital /ID# 78948, Kansas City, Missouri
  - Cardinal Glennon Children's Ho /ID# 79275, St Louis, Missouri
  - Children's Hospital St Louis /ID# 78910, St Louis, Missouri
  - Univ Nebraska Med Ctr /ID# 78932, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center /ID# 78957, Lebanon, New Hampshire
  - St. Barnabas Medical Center /ID# 79258, Livingston, New Jersey
  - Monmouth Medical Center /ID# 78901, Long Branch, New Jersey
  - Goryeb Chidlren's Hospital /ID# 76782, Morristown, New Jersey
  - Rutgers Robert Wood Johnson /ID# 119978, New Brunswick, New Jersey
  - Albany Medical College /ID# 76774, Albany, New York
  - Cystic Fibrosis Therapeutics /ID# 78941, Buffalo, New York
  - North Shore University Hospital /ID# 76779, New Hyde Park, New York
  - Mount Sinai Beth Israel /ID# 76773, New York, New York
  - Columbia Univ Medical Center /ID# 79376, New York, New York
  - Univ Rochester Med Ctr /ID# 92713, Rochester, New York
  - SUNY Upstate Medical University - Downtown /ID# 78912, Syracuse, New York
  - New York Medical College /ID# 78956, Valhalla, New York
  - Univ NC Chapel Hill /ID# 78937, Chapel Hill, North Carolina
  - Duke University Medical Center /ID# 79393, Durham, North Carolina
  - Mid Dakota Clinic, PC /ID# 78958, Bismarck, North Dakota
  - Akron Childrens Hospital /ID# 79263, Akron, Ohio
  - Cincinnati Children's Hospital /ID# 79375, Cincinnati, Ohio
  - University of Cincinnati /ID# 76789, Cincinnati, Ohio
  - Case Western Reserve Univ /ID# 78904, Cleveland, Ohio
  - Nationwide Childrens Hospital /ID# 78897, Columbus, Ohio
  - The Childrens Medical Center /ID# 78915, Dayton, Ohio
  - ProMedica Toledo Hospital /ID# 78913, Toledo, Ohio
  - Univ Oklahoma HSC /ID# 79279, Oklahoma City, Oklahoma
  - Kaiser Permanente, NW /ID# 79236, Portland, Oregon
  - Oregon Health and Science University /ID# 78900, Portland, Oregon
  - Geisinger Medical Center /ID# 79233, Danville, Pennsylvania
  - Penn State Child Hosp.Hersh,PA /ID# 79398, Hershey, Pennsylvania
  - Children's Hosp Philadelphia /ID# 79280, Philadelphia, Pennsylvania
  - Drexel Univ College of Med /ID# 76777, Philadelphia, Pennsylvania
  - St. Christopher's Hospital /ID# 78908, Philadelphia, Pennsylvania
  - Child Hosp of Pittsburgh,PA /ID# 79281, Pittsburgh, Pennsylvania
  - Rhode Island Hospital /ID# 79274, Providence, Rhode Island
  - Medical University of South Carolina /ID# 79262, Charleston, South Carolina
  - Sanford Research/USD /ID# 78909, Sioux Falls, South Dakota
  - LeBonheur Children's Med Ctr /ID# 78938, Memphis, Tennessee
  - Vanderbilt Univ Med Ctr /ID# 78947, Nashville, Tennessee
  - Specially for Children /ID# 79213, Austin, Texas
  - UT Southwestern Medical Center /ID# 78914, Dallas, Texas
  - Cook Children's Med. Center /ID# 78949, Fort Worth, Texas
  - Baylor College of Medicine /ID# 79273, Houston, Texas
  - Univ Texas HSC San Antonio /ID# 79374, San Antonio, Texas
  - The Univ Texas HSC at Tyler /ID# 79261, Tyler, Texas
  - University of Utah /ID# 76794, Salt Lake City, Utah
  - University of Vermont Medical Center /ID# 78933, Burlington, Vermont
  - University of Virginia /ID# 78942, Charlottesville, Virginia
  - Child Hosp of the King's Dtr's /ID# 79293, Norfolk, Virginia
  - Children's Hospital of Richmon /ID# 78955, Richmond, Virginia
  - Seattle Children's Hospital /ID# 78902, Seattle, Washington
  - Arthritis Northwest, PLLC /ID# 79257, Spokane, Washington
  - West Virginia Univ School Med /ID# 78953, Morgantown, West Virginia
  - Univ of Wisconsin Hosp/Clinics /ID# 78944, Madison, Wisconsin
  - Froedtert & the Medical College of Wisconsin /ID# 76778, Milwaukee, Wisconsin
  - Children's Hospital Wisconsin - Milwaukee Campus /ID# 79294, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chiuve SE, Fife D, Leitz G, Peterson C, Campbell NM, Rennig A, Rodrigues L Jr, Decktor D, Dowd C, Marshall BC, Borowitz D. Incidence of fibrosing colonopathy with pancreatic enzyme replacement therapy in patients with cystic fibrosis. J Cyst Fibros. 2023 Nov;22(6):1017-1023. doi: 10.1016/j.jcf.2023.08.013. Epub 2023 Oct 23. PMID 37880023
- See also: clinical study report synopsis — https://www.abbvie.com/content/dam/abbvie-dotcom/clinical-trials/pancrelipase_CFFC-OB-11.pdf